CLINICAL TRIAL: NCT04768114
Title: Toward the Implementation of Genomics in Substance Use Disorder Treatment
Brief Title: Implementation of Genomics in Substance Use Disorder Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201704049; K12DA041449 (NIH)
Record Dates: First submitted 2021-02-11; First posted 2021-02-24 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Tobacco Use Disorder; Smoking Cessation; Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genetically-Informed RiskProfile (Experimental)
  Interventions: Behavioral: Genetically-Informed RiskProfile
- Brief Cessation Advice (Active Comparator)
  Interventions: Other: Brief Cessation Advice

INTERVENTIONS:
Behavioral: Genetically-Informed RiskProfile — * Participants will meet with a behavioral interventionist to receive their personalized genetically-informed RiskProfile intervention which incorporates smoking-related genetic risk propensity and phenotypic risk (cigarettes smoked per day) into a risk communication tool designed to activate behavior change, specifically, to increase the use of smoking cessation medications and promote smoking-related behavior change.
  * This is a fully remote trial, with intervention delivered via video conferencing.
  Arms: Genetically-Informed RiskProfile
Other: Brief Cessation Advice — * Participants will meet with a behavioral interventionist to receive standardized brief advice to quit smoking and encouragement to use freely-available smoking cessation resources. Participants will receive their personalized RiskProfile after all data collection has been completed.
  * This is a fully remote trial, with brief cessation advice delivered via video conferencing.
  Arms: Brief Cessation Advice

SUMMARY:
Cigarette smoking remains one of the leading causes of preventable death. Effective smoking cessation medications exist but use of these treatments is low, making it difficult for most to quit smoking. Behavioral interventions are needed to engage current smokers in the process of quitting smoking and promote the use of evidence-based cessation medications.

At the same time, genetics influences one's smoking behaviors (e.g., how much they smoke, difficulty quitting) and risk of smoking-related diseases, yet these personalized factors have not been included in existing behavioral interventions. Incorporating these individualized factors into smoking cessation interventions may make them more personally engaging and thus motivating for treatment.

This study will pilot test a risk communication tool that is personalized to one's genetics and will demonstrate the feasibility of a larger trial to test the effect of this personalized genetically-informed intervention on smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Smoked combustible cigarettes in past 30 days
* Computer access for remote-based study visits

Exclusion Criteria:

* Younger than 18 years of age
* No computer access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex T Ramsey, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
* Project data will be shared in de-identified form in accordance with NIH policies including the NIH Genomic Data Sharing Policy. The informed consent process will explain policies for sharing de-identified data with other investigators and NIH repositories.
  * Even though the dataset to be shared will be stripped of identifiers prior to release for sharing, there may be the possibility of deductive disclosure of subjects with unusual characteristics. Thus, the investigators will make the individual-level data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to use the data only for research purposes and not attempt to identify any individual participant; (2) a commitment to store the data on a secure server and take necessary precautions to protect the security of the data; and (3) a commitment to destroy the data after analyses are completed.
Time Frame: Plan to publish within 12 months of ending data collection.
Access Criteria: The investigators will disseminate study findings through manuscripts, presentations, and lay reports. The investigators will make available via publications the steps and programs needed to implement the intervention. The investigators will make the protocols and tools available to other researchers to be used as a model template for interventions bringing genetics to the treatment of other substance use disorders.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 02/08/2021 and closed to participant enrollment on 05/29/2022.
Groups:
- Genetically-Informed RiskProfile: Participants will meet with a behavioral interventionist to receive their personalized genetically-informed RiskProfile intervention which incorporates smoking-related genetic risk propensity and phenotypic risk (cigarettes smoked per day) into a risk communication tool designed to activate behavior change, specifically, to increase the use of smoking cessation medications and promote smoking-related behavior change.
  This is a fully remote trial, with intervention delivered via video conferencing.
- Brief Cessation Advice: Participants will meet with a behavioral interventionist to receive standardized brief advice to quit smoking and encouragement to use freely-available smoking cessation resources. Participants will receive their personalized RiskProfile after all data collection has been completed.
  This is a fully remote trial, with brief cessation advice delivered via video conferencing.
Period: Overall Study
Arm/Group | Genetically-Informed RiskProfile | Brief Cessation Advice
Started | 74 | 74
Completed | 69 | 63
Not Completed | 5 | 11
Not completed — Lost to Follow-up | 5 | 10
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genetically-Informed RiskProfile | Brief Cessation Advice | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 68 | 62 | 130
  >=65 years | 6 | 12 | 18
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 51 | 54 | 105
  Male | 21 | 19 | 40
  Trans female / trans w | 0 | 1 | 1
  Non-binary | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 73 | 74 | 147
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 25 | 52
  White | 45 | 45 | 90
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 74 | 74 | 148

OUTCOME MEASURES:

1. Primary Outcome: Change in Use of Smoking Cessation Pharmacotherapy in Past 30 Days
Description: Participants in both groups were asked about their use of several smoking cessation medications (Question: "In the past 30 days, have you used any of the following prescription medications or over-the-counter aids to help you quit or cut back on smoking?"; Response options: 1=Bupropion or Zyban; 2=Varenicline or Chantix; 3=Nicotine patch; 4=Nicotine gum or lozenge; 5=Other (Specify).
Time Frame: Baseline, immediately prior to intervention receipt, 30-day follow-up, and 6-month follow-up
Population: Some participants did not complete assessments at prior to intervention, 30-day follow-up and 6 month follow-up so that is why the number of participants analyzed at these time points does not match the number of participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Genetically-Informed RiskProfile | Brief Cessation Advice
Number analyzed (Participants) | 74 | 74
Participants
  Self-reported use of any smoking cessation medications at baseline | 11 | 9
  Self-reported use of any smoking cessation medications at prior to intervention: number analyzed (Participants) | 72 | 66
  Self-reported use of any smoking cessation medications at prior to intervention | 9 | 2
  Self-reported use of any smoking cessation medications at 30-day follow-up: number analyzed (Participants) | 71 | 65
  Self-reported use of any smoking cessation medications at 30-day follow-up | 16 | 8
  Self-reported use of any smoking cessation medications at 6-month follow-up: number analyzed (Participants) | 69 | 63
  Self-reported use of any smoking cessation medications at 6-month follow-up | 15 | 8

2. Primary Outcome: Change in Number of Cigarettes Smoked Per Day
Description: Participants in both groups were asked "In the past 30 days, how many days did you smoke cigarettes" and "On the days in which you smoked cigarettes in the past month, about how many cigarettes did you smoke". The values from these questions are multiplied together and then divided by 30 (days) to calculate the number of cigarettes smoked per day for each participant.
Time Frame: Baseline, immediately prior to intervention receipt, 30-day follow-up, and 6-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cigarettes smoked per day
Arm/Group | Genetically-Informed RiskProfile | Brief Cessation Advice
Number analyzed (Participants) | 74 | 74
cigarettes smoked per day
  Self-reported cigarettes per day at baseline | 13.1 (8.2) | 12.3 (7.7)
  Self-reported cigarettes per day at prior to intervention: number analyzed (Participants) | 72 | 66
  Self-reported cigarettes per day at prior to intervention | 12.0 (8.5) | 11.5 (7.5)
  Self-reported cigarettes per day at 30-day follow-up: number analyzed (Participants) | 71 | 65
  Self-reported cigarettes per day at 30-day follow-up | 9.2 (8.4) | 9.7 (7.5)
  Self-reported cigarettes per day at 6-month follow-up: number analyzed (Participants) | 69 | 63
  Self-reported cigarettes per day at 6-month follow-up | 7.3 (7.3) | 9.1 (8.1)

3. Secondary Outcome: Change in Readiness to Quit Smoking
Description: Participants in both groups were assessed on self-reported stage of readiness to quit smoking.
  This measure includes one item based on the Transtheoretical Model of Change and measured along stages of Precontemplation, Contemplation, Preparation, and Action. (Question: ""Are you thinking of quitting smoking?""; Response options: 1=No, I am not seriously considering quitting within the next 6 months (Precontemplation); 2=Yes, I am seriously considering quitting within the next 6 months (Contemplation); 3=Yes, I am seriously planning to quit within the next 30 days (Preparation); 4=I have quit smoking within the past 6 months (Action). A higher score represents a higher stage of readiness to quit smoking. "
Time Frame: Baseline, immediately prior to intervention receipt, 30-day follow-up, and 6-month follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Genetically-Informed RiskProfile | Brief Cessation Advice
Number analyzed (Participants) | 74 | 74
Participants
  Baseline, Precontemplation count | 16 | 22
  Baseline, Contemplation count | 45 | 37
  Baseline, Preparation count | 13 | 15
  Baseline, Action count | 0 | 0
  Prior to intervention, Precontemplation count: number analyzed (Participants) | 71 | 66
  Prior to intervention, Precontemplation count | 12 | 13
  Prior to intervention, Contemplation count: number analyzed (Participants) | 71 | 66
  Prior to intervention, Contemplation count | 41 | 39
  Prior to intervention, Preparation count: number analyzed (Participants) | 71 | 66
  Prior to intervention, Preparation count | 17 | 13
  Prior to intervention, Action count: number analyzed (Participants) | 71 | 66
  Prior to intervention, Action count | 1 | 1
  30-day follow-up, Precontemplation count: number analyzed (Participants) | 71 | 65
  30-day follow-up, Precontemplation count | 8 | 12
  30-day follow-up, Contemplation count: number analyzed (Participants) | 71 | 65
  30-day follow-up, Contemplation count | 37 | 36
  30-day follow-up, Preparation count: number analyzed (Participants) | 71 | 65
  30-day follow-up, Preparation count | 22 | 13
  30-day follow-up, Action count: number analyzed (Participants) | 71 | 65
  30-day follow-up, Action count | 4 | 4
  6-month follow-up, Precontemplation count: number analyzed (Participants) | 68 | 63
  6-month follow-up, Precontemplation count | 13 | 4
  6-month follow-up, Contemplation count: number analyzed (Participants) | 68 | 63
  6-month follow-up, Contemplation count | 29 | 43
  6-month follow-up, Preparation count: number analyzed (Participants) | 68 | 63
  6-month follow-up, Preparation count | 16 | 9
  6-month follow-up, Action count: number analyzed (Participants) | 68 | 63
  6-month follow-up, Action count | 10 | 7

4. Secondary Outcome: Change in Perceived Disease Risk
Description: Participants in both groups were assessed on self-reported perceptions of personal susceptibility to smoking-related diseases. This measure includes one item comprising the perceived susceptibility scale (Question: "How likely is it for you to develop a smoking-related disease such as lung cancer or chronic obstructive pulmonary disease (COPD), if you continue to smoke?"; Response options: 1=Very unlikely; 2=Somewhat unlikely; 3=Neither unlikely nor likely; 4=Somewhat likely; 5=Very likely). A higher score represents a higher perceived disease risk.
Time Frame: Baseline, immediately following intervention receipt, 30-day follow-up, and 6-month follow-up
Population: Some participants did not complete assessments at baseline, immediately following intervention, 30-day follow-up and 6 month follow-up so that is why the number of participants analyzed at these time points does not match the number of participants enrolled.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genetically-Informed RiskProfile | Brief Cessation Advice
Number analyzed (Participants) | 72 | 72
score on a scale
  Baseline | 4.5 (0.8) | 4.3 (0.8)
  Immediately following intervention receipt: number analyzed (Participants) | 72 | 66
  Immediately following intervention receipt | 4.7 (0.7) | 4.3 (1.0)
  30-day follow-up: number analyzed (Participants) | 72 | 65
  30-day follow-up | 4.6 (0.6) | 4.4 (0.8)
  6-month follow-up: number analyzed (Participants) | 69 | 63
  6-month follow-up | 4.6 (0.8) | 4.5 (0.8)

5. Secondary Outcome: Change in Perceived Benefits of Cessation
Description: Participants in both groups were assessed on self-reported perceptions of personal health benefits related to quitting smoking. This measure is based on 3 items from the Perceived Risks and Benefits Questionnaire (PRBQ) addressing benefits related to reduced risks of smoking-related diseases, avoidance of future health problems, and increased longevity if the participant were to quit smoking. Response options to individual items were assessed on a 5-point Likert-type scale ranging from 1=Very Unlikely to 5=Very Likely. Individual scores on the 3 items were then averaged together for a total scale range of 1 to 5. A higher score represents higher perceived benefits of cessation.
Time Frame: Baseline, immediately following intervention receipt, 30-day follow-up, and 6-month follow-up
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genetically-Informed RiskProfile | Brief Cessation Advice
Number analyzed (Participants) | 74 | 73
score on a scale
  Self-reported perception of benefits of cessation at baseline | 4.2 (0.8) | 4.2 (0.8)
  Self-reported perception of benefits of cessation immediately following intervention receipt: number analyzed (Participants) | 72 | 66
  Self-reported perception of benefits of cessation immediately following intervention receipt | 4.2 (1.0) | 4.2 (0.8)
  Self-reported perception of benefits of cessation at 30-day follow-up: number analyzed (Participants) | 71 | 65
  Self-reported perception of benefits of cessation at 30-day follow-up | 4.6 (0.7) | 4.4 (0.7)
  Self-reported perception of benefits of cessation at 6-month follow-up: number analyzed (Participants) | 69 | 63
  Self-reported perception of benefits of cessation at 6-month follow-up | 4.6 (0.6) | 4.4 (0.7)

6. Secondary Outcome: Change in Perceived Value of Cessation Treatments
Description: Participants in both groups were assessed on self-reported perceptions of the importance of using smoking cessation medications to help quit smoking.
  This measure includes 4 items modified from the Beliefs and Attitudes about Buproprion Scale which assesses perceived importance of using medications for smoking cessation, perceived confidence in medications as a smoking cessation aid, general expectancy that smoking cessation medications help people stop smoking, and perceived confidence in being able to use smoking cessation medications within the next month. Response options to individual items were assessed on a 5-point Likert-type scale ranging from 1=Not at all to 5=Extremely. Individual scores on the 4 items were then averaged together for at total scale range of 1-5. A higher score represents a higher perceived value of cessation treatment.
Time Frame: Baseline, immediately following intervention receipt, 30-day follow-up, and 6-month follow-up
Population: Some participants did not complete assessments at immediately following intervention, 30-day follow-up and 6 month follow-up so that is why the number of participants analyzed at these time points does not match the number of participants enrolled.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genetically-Informed RiskProfile | Brief Cessation Advice
Number analyzed (Participants) | 74 | 74
score on a scale
  Baseline | 3.0 (0.9) | 3.0 (0.9)
  Immediately following intervention receipt: number analyzed (Participants) | 72 | 66
  Immediately following intervention receipt | 3.3 (0.9) | 2.9 (0.8)
  30-day follow-up: number analyzed (Participants) | 71 | 65
  30-day follow-up | 3.2 (1.0) | 2.9 (0.9)
  6-month follow-up: number analyzed (Participants) | 69 | 63
  6-month follow-up | 3.0 (1.1) | 2.8 (1.0)

7. Secondary Outcome: Change in Self-efficacy of Cessation
Description: Participants in both groups were assessed on self-reported perceptions of personal ability to engage in activities that promote smoking cessation. This measure is based on 3 items modified from the Skill Self-Efficacy Scale and 3 items modified from the Try Self-Efficacy Scale. Skill self-efficacy items address confidence to solicit social support, avoid situations with a high risk of relapse, and distract oneself when experiencing cravings during a quit attempt. Try self-efficacy items address perceived personal ability to smoke fewer cigarettes a day, resist smoking for one week, and resist smoking for one month. Response options to individual items were assessed on a 5-point Likert-type scale ranging from 1=Not at all to 5=Very. Individual scores on the 3 items were then averaged together for a total scale range of 1-5. A higher score represents a higher perceived self-efficacy of cessation.
Time Frame: Baseline, immediately following intervention receipt, 30-day follow-up, and 6-month follow-up
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genetically-Informed RiskProfile | Brief Cessation Advice
Number analyzed (Participants) | 74 | 74
score on a scale
  Self-reported skill self-efficacy at baseline | 3.5 (0.9) | 3.5 (0.8)
  Self-reported skill self-efficacy immediately following intervention receipt: number analyzed (Participants) | 72 | 66
  Self-reported skill self-efficacy immediately following intervention receipt | 3.6 (0.7) | 3.7 (0.7)
  Self-reported skill self-efficacy at 30-day follow-up: number analyzed (Participants) | 71 | 65
  Self-reported skill self-efficacy at 30-day follow-up | 3.8 (1.0) | 3.9 (0.8)
  Self-reported skill self-efficacy at 6-month follow-up: number analyzed (Participants) | 69 | 63
  Self-reported skill self-efficacy at 6-month follow-up | 3.9 (1.0) | 3.9 (0.9)
  Self-reported try self-efficacy at baseline | 2.6 (1.0) | 2.6 (1.0)
  Self-reported try self-efficacy immediately following intervention receipt: number analyzed (Participants) | 72 | 66
  Self-reported try self-efficacy immediately following intervention receipt | 2.6 (1.0) | 2.6 (1.0)
  Self-reported try self-efficacy at 30-day follow-up: number analyzed (Participants) | 71 | 65
  Self-reported try self-efficacy at 30-day follow-up | 2.8 (1.2) | 3.0 (1.1)
  Self-reported try self-efficacy at 6-month follow-up: number analyzed (Participants) | 69 | 63
  Self-reported try self-efficacy at 6-month follow-up | 3.2 (1.4) | 3.4 (1.2)

8. Secondary Outcome: Personal Relevance of Intervention
Description: Participants in both groups were assessed on self-reported perceptions of the extent to which the intervention was personally significant and applicable. This measure includes 4 items modified from the Personal Relevance Scale and addresses the extent to which the intervention helped participants learn something about themselves, the role that their personal characteristics play in their smoking, how smoking affects their life, and the impact on their smoking cessation attempts. Response options to individual items were assessed on a 5-point Likert-type scale ranging from 1=Strongly Disagree to 5=Strongly Agree. Individual scores on the 4 items were then averaged together for a total scale range of 1 to 5. A higher score represents a higher perception of personal relevance of the intervention.
Time Frame: Immediately following intervention receipt
Population: Some participants did not complete the assessment immediately following intervention so that is why the number of participants analyzed does not match the number of participants enrolled.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genetically-Informed RiskProfile | Brief Cessation Advice
Number analyzed (Participants) | 72 | 66
score on a scale | 4.5 (0.6) | 3.7 (0.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at baseline, immediately following intervention receipt, 30-day follow-up, and 6-month follow-up.
Description: Adverse events were collected when self-reported by participants during the trial.
Arm/Group | Genetically-Informed RiskProfile | Brief Cessation Advice
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74
Other Adverse Events (participants affected / at risk) | 1/74 | 0/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genetically-Informed RiskProfile (N=74) | Brief Cessation Advice (N=74)
Anxiety (Psychiatric disorders) | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT04768114/Prot_SAP_000.pdf